CLINICAL TRIAL: NCT01054274
Title: Self-Expandable Esophageal Radiation Stent:a Multicentric Randomized Controlled Trial in Patients With Advanced Esophageal Cancer
Brief Title: a Multicentric Randomized Controlled Trial of Self-Expandable Esophageal Radiation Stent
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Gao-Jun Teng, Director, Southeast University, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 320924197612177170
Record Dates: First submitted 2010-01-21; First posted 2010-01-22 (Estimated); Last update posted 2012-04-02 (Estimated); Status verified 2009-12

CONDITIONS: Esophageal Cancer
Keywords: esophageal cancer; dysphagia; stent; brachytherapy
MeSH Terms: conditions — Esophageal Neoplasms; Deglutition Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- novel stent (Active Comparator): Patients undergo placement of a novel esophageal stent loaded with 125I seeds on day 1.
  Interventions: Device: novel stent
- conventional covered stent (Experimental): Patients undergo placement of a conventional covered stent on day 1.
  Interventions: Device: conventional covered stent

INTERVENTIONS:
Device: novel stent — Patients undergo placement of a novel esophageal stent loaded with 125I seeds on day 1.
  Other Names: self-expandable esophageal radiation stent
  Arms: novel stent
Device: conventional covered stent — Patients undergo placement of a conventional covered stent on day 1.
  Other Names: conventional stent
  Arms: conventional covered stent

SUMMARY:
Esophageal cancer is common in some areas , ranking as the fourth leading cause of death from cancer in China and sixth worldwide. Although the prognosis of surgical resection for esophageal cancer has been improved, more than 50% of such patients are inoperable and have to undergo palliative treatments because of late stage cancer or metastasis. Dysphagia is the predominate symptom of patients with inoperable esophageal cancer. To relieve the dysphagia and improve the quality of life of such patients, brachytherapy has previously been utilized. Recently, stent placement has been widely accepted to be an option for palliation of the symptoms due to the esophageal strictures. Brachytherapy and esophageal self-expanding stent insertion have longer benefit. Stent insertion provides fastest improvement of dysphagia.However, recurrence of the neoplastic stricture remains a challenge after stent placement, complications in later setting occur and require further endoscopic treatment. Brachytherapy has slower onset of benefit but has fewer complications and longer benefit.To combine the advantages of the immediate relief of the esophageal dysphagia with the stent placement and radiation therapy with brachytherapy, a novel esophageal stent loaded with 125I seeds has been developed in the authors' institute. The technical feasibility and safety with this new stent has been demonstrated to be adequate in a healthy rabbit model. And a small-sample and unicentric prior clinical trial in the authors' institute certificated the novel esophageal stent can relieve the dysphagia caused by advanced esophageal cancer rapidly and improve the quality of life markedly. This current multicentric randomized clinical trial is further studying the novel esophageal stent loaded with 125I seeds to see how well they work compared with a conventional covered stent in patients with malignant dysphagia caused by advanced esophageal cancer.

DETAILED DESCRIPTION:
PURPOSE Rationale: Placing a stent in the esophagus may relieve the dysphagia caused by inoperable esophageal cancer rapidly and improve the quality of life . But recurrence of the neoplastic stricture remains a challenge after solitary stent placement. Brachytherapy is an option for palliation of the symptoms due to the esophageal strictures,however,it can not relieve the dysphagia rapidly. So a novel esophageal stent loaded with 125I seeds combines the advantages of the immediate relief of the esophageal dysphagia with the stent placement and radiation therapy with brachytherapy.

Purpose: A small-sample and unicentric clinical trial in the authors' institute had certificated that a novel esophageal stent loaded with 125I seeds for intraluminal brachytherapy can relieve the dysphagia caused by advanced esophageal cancer rapidly and improve the quality of life . This multicentric randomized clinical trial is further studying the novel esophageal stent loaded with 125I seeds to see how well they work compared with a conventional covered stent in patients with malignant dysphagia caused by advanced esophageal cancer.

OUTLINE: This is a multicentric, randomized, controlled study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo placement of a novel esophageal stent loaded with 125I seeds on day 1.
* Arm II: Patients undergo placement of a conventional covered stent on day 1.
* Health-related quality of life is assessed at baseline, I, 3 and 6 months.

Condition :Esophageal Cancer Intervention (Procedure): Esophageal stent placement,dysphagia scores,complications of therapy,survival time of therapy Phase :Ⅲ

DISEASE AND PATIENT CHARACTERISTICS:

Criteria

Inclusion Criteria:

* Endoscopically and histologically confirmed cancer of esophagus,
* Progressive dysphagia caused by esophageal cancer, and the dysphagia grade of level Ⅲ or level Ⅳ[STOOLER stand],
* In barium meal of esophagus, severe stricture of the cancer make the barium difficult to pass through and the superior normal esophagus broaden,
* The bulk and shape of the oesophageal cancer displayed by CT three-dimensional reconstruction,
* Patients with clear consciousness，Cooperation，ECOG performance status of 0,1 and 3,
* Informed consent: authorization and signature.

Exclusion Criteria:

* Poor general status,ECOG performance status of 4,
* Dysphagia not caused by esophageal cancer,
* Noncooperation or no authorization and signature.
* The superior border of cancer higher than the seventh cervical vertebrae
* Ulcerative esophageal carcinoma
* Esophageal fistulas,
* WBC less than 3000/mm3
* Severe hepatic inadequacy or renal inadequacy,

Exit or Termination Criteria:

Patient Exit :

* Patient who ask to exit actively,
* Patient who can not collaborate with relative tests and effect the date collection,
* Receiving other therapies without permission, such as, chemotherapy,radiotherapy, etc.,
* Occurring of other disease or severe complications simultaneously make the patient need to be rescued immediately and will effect the trial.

Termination:

* Severe safety questions,such as the follow-up death after the stent insertion,
* Severe lapsus of the trial design leads ro difficulty in efficacy evaluation about stent,
* Severe bias in the practice of trial leads ro difficulty in efficacy evaluation about equipment.

Case exfoliation :

Definition:any participant who has signed and entered the trial do not insist to the end.The reasons may be:

* The participant do not cooperate with the designed tests or receive other therapies without the permission,
* The participant exfoliate from the trial or follow-up lost ,
* Severe adverse reactions,events or complications make the participant can not keep on the treatment.

Exfoliation handle:

* Inquest the reason and supply the date by telephone and follow-up visiting,
* Corresponding methods should be adapted to handle the adverse reactions,adverse events or complications,
* Store the primitive date of exfoliated participants for full analysis set（FAS）statistics.

Case rejection:

* Misdiagnosis and wrong enrollment,
* Consistent with exclusion criteria,
* No any test record,
* Can not evaluate the efficacy for receiving other therapies without the permission, Any rejected case should be supplied with the reason and quit the curative effect statistical analysis.However, the record of those who have been treated for at least one time should be included into the adverse reactions analysis.

RANDOMIZATION

Trial design:

* Multicentre: all patients come from sixteen hospitals disseminated in China,
* Completely randomized：Number are completely randomized formed depending on the SAS statistics software and are administered by the sponsor,every collaborator apply for the number once a participant enrolled and choose the treatment arm according to the random number.
* Single Blind:the participants is unaware which treatment will to be took
* Active Control: there are treatment arms. Arm I: patients undergo placement of a novel esophageal stent loaded with 125I seeds. Arm II: patients undergo placement of a conventional covered stent.
* Sample estimation:It has been demonstrated in the preclinical trial that the median survival time of the advanced esophageal cancer patients with self-expandable esophageal radiation stent insertion is about 7 m, while those with conventional covered stent insertion is about 4 m. Considering the enrollment time of 3 m(T1 is 0.25y),whole trial time of 1.5y.and α is 0.05 (test of two-sided) or 0.10(test of one-sided），the least sample number is 152.If the exfoliated cases are considered, the least sample number is 186 (increasing about 20 percent).

Case diffusion

Be sent to one of two arms according to the random number randomized formed by the SAS statistics software.

Radiation dose estimation:

After balloon dilation ( the special balloon producted for esophageal dilation by Nanjing MicroInvasive Medical,Nanjing,China) in participants[the balloon diameter is 16mm in superior segment of esophagus and 18mm in the midpiece and inferior segment of esophagus],CT scan of the esophagus with the balloon in is performed.Then the images will be send to the Treatment Planning System(TPS, Nanjing MicroInvasive Medical,Nanjing,China),and the bulk of the oesophageal cancer will be calculated according to the CT three-dimensional reconstruction images.At last,the radiation dose will be estimated(with radioactivity 0.7mCi according to the preclinical study).

Choice of stent and seeds fixation:

The esophageal irradiation stent combined a self-expandable covered esophageal stent(MTN;Nanjing MicroInvasive Medical,Nanjing,China) loaded (or not loaded) with 125I radiative seeds(CIAE-6711;Chinese Atomic Energy Science Institution,Beijing,China) are chose.The diameter varies from 16 to 18mm(16mm in superior segment of esophagus and 18mm in the midpiece and inferior segment of esophagus), the length is the length of disease with additional 20mm. The seeds (number is decided according to the radiation dose estimated in advance)are fixed around the stent,covering the superior and inferior border of the cancer (the distance of seeds varies from 10mm to 15mm and the distance of seeds and inlet/outlet less than10mm).

Post-operation Care Participants lie on the back with waist raised after stent insertion, common treatments include hemostasis, infection prevention, mucous membrane of esophagus and stomach protection.No cold diet,except eating fluid slowly.

Follow-up

Calling or visiting the patients every month after test insertion.

Objectives:

[Time Frame: Follow-up in intervals of 1, 3, 6, and 12 months after stent placement ]

Primary:

* Overall survival
* Median Survival

Secondary

* Quality of life [ECOG performance status]
* Dysphagia grade [STOOLER stand]
* Change of the oesophageal cancer [ RECIST standard]
* Restenosis degree[esophagus visualization]
* Pathologic change of the cancer,
* Successful rate of stent placement,

Safety

* Immune function(IgA,IgG,IgM,CD3,CD4,CD4/CD8)
* Myelosuppression
* Distribution and attenuation of isotope[ECT or PET]
* Adverse events [CTCAE v3.0 standard] Determine the individual rates of complication associated with each type of esophageal stent in these patients.

Statistical analysis:

All primal date should be stored completely and precisely and submitted to the special date administrator in time by the Internet.Before entering the date into the special database by two people independent, all submitted data must be reviewed, verified to ensure the accuracy, currency(according to the primal date).

Statistical analysis software of SAS 9.0 is adapted. Test of two-sided, if P ≤0.05,there are significant difference. Mean, standard deviation(SD),median, maximum and minimum value are used to describe the measurement data of two groups;the rank sum test is used to valuate the relief of dysphagia;log-rank test is used to compare the survival curves of two groups which have been drawn with the Kaplan-meier method.At last the median survivals will be obtained and compared by t test and rank sum test .

Constituent ratio is used to describe the numeration data of two groups; u test is used to valuate the difference of survival rates;and the reasons of restenosis are analysed with Fisher's exact test or chi-square(X2) test.

The balance-analyses of fundament data(population data and others): t test or chi-square(X2) test is chose.

Esophageal Cancer PURPOSE Rationale: Placing a stent in the esophagus may relieve the dysphagia caused by inoperable esophageal cancer rapidly and improve the quality of life . But recurrence of the neoplastic stricture remains a challenge after solitary stent placement. Brachytherapy is an option for palliation of the symptoms due to the esophageal strictures,however,it can not relieve the dysphagia rapidly. So a novel esophageal stent loaded with 125I seeds combines the advantages of the immediate relief of the esophageal dysphagia with the stent placement and radiation therapy with brachytherapy.

Purpose: A small-sample and unicentric clinical trial in the authors' institute had certificated that a novel esophageal stent loaded with 125I seeds for intraluminal brachytherapy can relieve the dysphagia caused by advanced esophageal cancer rapidly and improve the quality of life . This multicentric randomized clinical trial is further studying the novel esophageal stent loaded with 125I seeds to see how well they work com

ELIGIBILITY:
Inclusion Criteria:

* Endoscopically and histologically confirmed cancer of esophagus
* Progressive dysphagia caused by esophageal cancer, and the dysphagia grade of level Ⅲ or level Ⅳ[STOOLER stand]
* In barium meal of esophagus, severe stricture of the cancer make the barium difficult to pass through and the superior normal esophagus broaden
* The bulk and shape of the oesophageal cancer displayed by CT three-dimensional reconstruction
* Patients with clear consciousness，Cooperation，ECOG performance status of 0,1 and 3
* Informed consent: authorization and signature

Exclusion Criteria:

* Poor general status,ECOG performance status of 4,
* Dysphagia not caused by esophageal cancer,
* Noncooperation or no authorization and signature.
* The superior border of cancer higher than the seventh cervical vertebrae
* Ulcerative esophageal carcinoma
* Esophageal fistulas,
* WBC less than 3000/mm3

  * Severe hepatic inadequacy or renal inadequacy,

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2009-12; Primary Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival and Median Survival | Follow-up in intervals of 1, 3, 6, and 12 months after stent placement

SECONDARY OUTCOMES:
Quality of life [ECOG performance status],Dysphagia grade [STOOLER stand],Change of the oesophageal cancer [ RECIST standard],Restenosis degree[esophagus visualization] | Follow-up in intervals of 1, 3, 6, and 12 months after stent placement
Pathologic change of the cancer | Follow-up in intervals of 1, 3, 6, and 12 months after stent placement
Successful rate of stent placement | Follow-up in intervals of 1, 3, 6, and 12 months after stent placement

CONTACTS AND LOCATIONS:
Overall Officials: Gao-Jun Teng, MD, Principal Investigator — Medical School,Southeast University
Locations (1):
- Zhongda Hospital, Southeast University, Nanjing, Jiangsu, China

REFERENCES:
- [Result] Guo JH, Teng GJ, Zhu GY, He SC, Deng G, He J. Self-expandable stent loaded with 125I seeds: feasibility and safety in a rabbit model. Eur J Radiol. 2007 Feb;61(2):356-61. doi: 10.1016/j.ejrad.2006.10.003. Epub 2006 Nov 7. PMID 17085003
- [Result] Guo JH, Teng GJ, Zhu GY, He SC, Fang W, Deng G, Li GZ. Self-expandable esophageal stent loaded with 125I seeds: initial experience in patients with advanced esophageal cancer. Radiology. 2008 May;247(2):574-81. doi: 10.1148/radiol.2472070999. Epub 2008 Mar 18. PMID 18349316
- [Derived] Zhu HD, Guo JH, Mao AW, Lv WF, Ji JS, Wang WH, Lv B, Yang RM, Wu W, Ni CF, Min J, Zhu GY, Chen L, Zhu ML, Dai ZY, Liu PF, Gu JP, Ren WX, Shi RH, Xu GF, He SC, Deng G, Teng GJ. Conventional stents versus stents loaded with (125)iodine seeds for the treatment of unresectable oesophageal cancer: a multicentre, randomised phase 3 trial. Lancet Oncol. 2014 May;15(6):612-9. doi: 10.1016/S1470-2045(14)70131-7. Epub 2014 Apr 14. PMID 24742740